CLINICAL TRIAL: NCT01960725
Title: An Open-label, Pilot Study to Compare the Safety and Immunogenicity of an Alternate Dosing Schedule (2-5 Weeks, 2 Months, and 4 Months) for Pentavalent Rotavirus Vaccine (RotaTeq) to the Standard Recommended Schedule (2, 4, and 6 Months)
Brief Title: An Alternate Dosing Schedule for Pentavalent Rotavirus Vaccine (RotaTeq)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dennis Clements (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Dennis Clements, Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00049081; MISP-50891 (Other Grant/Funding Number: Merck Investigator Studies Program)
Record Dates: First submitted 2013-10-07; First posted 2013-10-11 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: Diarrhea; Gastroenteritis
Keywords: Gastroenteritis; Diarrhea; Rotavirus; Vaccine; Dehydration
MeSH Terms: conditions — Diarrhea; Gastroenteritis; Dehydration | interventions — RotaTeq

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Dosing Group (Active Comparator): Group will receive RV5 vaccine at 2, 4, and 6 months of age
  Interventions: Biological: RV5 (Pentavalent Rotavirus Vaccine)
- Alternate Dosing Group (Experimental): Group will receive RV5 vaccine at 2-5 weeks, 2 and 4 months of age
  Interventions: Biological: RV5 (Pentavalent Rotavirus Vaccine)

INTERVENTIONS:
Biological: RV5 (Pentavalent Rotavirus Vaccine)
  Other Names: RotaTeq

SUMMARY:
This is a pilot study to assess the safety and immunogenicity of pentavalent rotavirus vaccine (RV5) when administered according to an alternate dosing schedule (2-5 weeks, 2 months and 4 months). In this interventional, open-label study, infants 2 through 5 weeks of age (14 to 41 days) will be enrolled and vaccinated with RV5 according to a 2-5 week, 2 and 4 month schedule and infants 2 months of age (56 to 83 days) will be vaccinated according to the standard recommended schedule (2, 4, and 6 months of age). Sera will be obtained from subjects one month following the final dose of vaccine and will be assayed for anti-rotavirus IgA and rotavirus neutralizing antibody responses against the G1, G2, G3, G4 and P[8] serotypes. Post dose 3 G1 serum-neutralizing antibody (SNA) geometric mean titers (GMTs) will be compared between children receiving pentavalent rotavirus vaccine (RV5) according to the alternate dosing schedule versus the standard recommended schedule. Likewise, post dose 3 G2, G3, G4 and P[8] SNA and serum rotavirus IgA GMTs will be compared between children receiving RV5 according to the alternate dosing schedule and the standard recommended schedule. The safety and tolerability of RV5 in children receiving vaccine according to the alternate dosing schedule will be described.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female infants who are 14 through 41 or 56 through 83 days of age at Visit 1 (Day of initial vaccination)
2. Parent / legal guardian has read and signed the informed consent document
3. Child and parent / legal guardian is available for the entire study period and can be reached by telephone
4. Healthy infant as determined by medical history and by a baseline physical examination
5. Infant weight at time of enrollment must exceed birth weight

Exclusion Criteria:

1. History of hypersensitivity to the vaccine or any component of the vaccine
2. History of Severe Combined Immunodeficiency Disease (SCID)
3. History of immunocompromise ( infant is known to be HIV positive, to have hypogammaglobulinemia or to have an underlying malignancy)
4. History of intussusception
5. Any clinically significant history of gastrointestinal disease including active acute gastrointestinal illness, chronic diarrhea, failure to thrive, congenital abdominal disorders, abdominal surgery or liver disease
6. Prior receipt of a rotavirus vaccine
7. Less than 37 weeks gestation
8. The subject has participated in a study with an experimental agent within one month of enrollment in the study or anticipated receipt of an experimental agent during participation in the study
9. Receipt of blood products within 4 weeks of study vaccination
10. Receipt of a live virus vaccine within 4 weeks of study vaccination or an inactivated vaccine within 2 weeks. Concomitant administration of routinely recommended vaccines is allowed. A dose of hepatitis B vaccine administered in the birthing hospital is permitted. Planned routine use of inactivated influenza vaccine for children over 6 months of age is permitted.
11. Acute illness within 48 hours of vaccination (axillary temperature of 100.4°F or higher, 3 or more grossly watery stools, vomiting). (Infants with stable unchanged gastroesophageal reflux may be enrolled).
12. Insufficient weight gain requiring future weight checks in addition to routine scheduled well child visits
13. The subject has any condition that the investigator believes would put the subject at an increased risk of injury or would render the subject unable to complete the trial or fulfill the requirements of the study protocol.
14. Household contact who is immunodeficient (any malignancies or otherwise immunocompromised, primary immunodeficiency, receiving immunosuppressive therapy)

Ages: 14 Days to 83 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis A Clements, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Standard Dosing: Group will receive RV5 vaccine at 2, 4, and 6 months of age
  RV5 (Pentavalent Rotavirus Vaccine)
- Group B: Alternate Dosing: Group will receive RV5 vaccine at 2-5 weeks, 2 and 4 months of age
  RV5 (Pentavalent Rotavirus Vaccine)
Period: Overall Study
Arm/Group | Group A: Standard Dosing | Group B: Alternate Dosing
Started | 33 | 33
Received First Vaccine | 33 | 33
Recieved Second Vaccine | 33 | 33
Received Third Vaccine | 32 | 32
Completed (Immunogenicity data completed) | 27 | 28
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 4 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — unable to obtain blood sample | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Standard Dosing | Group B: Alternate Dosing | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: days] | 63 (4.6) | 26.6 (7.3) | 44.8 (19.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 40
  Male | 14 | 12 | 26
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 2 | 2
  White | 24 | 27 | 51
  African American | 9 | 4 | 13
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 3 | 3 | 6
  Non-Hispanic | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: G1 Serum-neutralizing Antibody
Description: Post dose 3 G1 serum-neutralizing antibody (SNA) geometric mean titer (GMT)
Time Frame: 1 month following vaccine series completion
Population: The per protocol analysis population includes participants who met all inclusion and exclusion criteria, received all scheduled study vaccinations, and who contributed post-vaccination blood samples for testing for which valid results were reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group A: Standard Dosing | Group B: Alternate Dosing
Number analyzed (Participants) | 27 | 28
titers | 188 [117.9 to 299.7] | 184.5 [117 to 290.8]

2. Secondary Outcome: G2 Serum-neutralizing Antibody
Description: Post dose 3 G2 serum-neutralizing antibody(SNA) geometric mean titer (GMT)
Time Frame: 1 month following vaccine series completion
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group A: Standard Dosing | Group B: Alternate Dosing
Number analyzed (Participants) | 27 | 28
titers | 38.7 [25 to 59.9] | 33.1 [20.7 to 52.9]

3. Secondary Outcome: G3 Serum-neutralizing Antibody
Description: Post dose 3 G3 serum-neutralizing antibody(SNA) geometric mean titer (GMT)
Time Frame: 1 month following vaccine series completion
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group A: Standard Dosing | Group B: Alternate Dosing
Number analyzed (Participants) | 27 | 28
titers | 42.1 [27.5 to 64.6] | 27.3 [17.3 to 43.2]

4. Secondary Outcome: G4 Serum-neutralizing Antibody
Description: Post dose 3 G4 serum-neutralizing antibody(SNA) geometric mean titer (GMT)
Time Frame: 1 month following vaccine series completion
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group A: Standard Dosing | Group B: Alternate Dosing
Number analyzed (Participants) | 27 | 28
titers | 144.6 [105.1 to 198.8] | 66.5 [50.7 to 87.1]

5. Secondary Outcome: P1 Serum-neutralizing Antibody
Description: Post dose 3 P1 serum-neutralizing antibody(SNA) geometric mean titer (GMT)
Time Frame: 1 month following vaccine series completion
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group A: Standard Dosing | Group B: Alternate Dosing
Number analyzed (Participants) | 27 | 28
titers | 114.7 [77.51 to 169.6] | 136.5 [84.91 to 219.3]

6. Other Pre Specified Outcome: Serum Rotavirus Immunoglobulin A
Description: Post dose 3 serum rotavirus Immunoglobulin A geometric mean titer (GMT)
Time Frame: 1 month following vaccine series completion
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group A: Standard Dosing | Group B: Alternate Dosing
Number analyzed (Participants) | 27 | 28
titers | 318.3 [179.7 to 563.8] | 183.7 [93.37 to 361.6]

7. Other Pre Specified Outcome: Reactogenicity Assessment
Description: Proportions of subjects in each vaccine group reporting a reactogenicity event in the period following each dose and any dose of RV5 will be determined
Time Frame: 7 days after each dose, up to 10 months post-vaccination
Population: Proportions of subjects in each vaccine group reporting a reactogenicity event in the period following each dose and any does of RV5 will be determined
Measure: Number; unit: Proportion of participants
Arm/Group | Group A: Standard Dosing | Group B: Alternate Dosing
Number analyzed (Participants) | 33 | 33
Proportion of participants
  Fever | 0.06 | 0.03
  Vomiting | 0.15 | 0.24
  Diarrhea | 0.21 | 0.39

8. Other Pre Specified Outcome: Adverse Event Assessment
Description: Proportions of subjects in each vaccine group reporting an adverse event in the period following each dose and any dose of RV5 will be determined
Time Frame: 28 days after each dose, up to 10 months post-vaccination
Measure: Number; unit: Proportion of participants
Arm/Group | Group A: Standard Dosing | Group B: Alternate Dosing
Number analyzed (Participants) | 33 | 33
Proportion of participants
  Post dose 1 | 0.27 | 0.51
  Post dose 2 | 0.06 | 0.09
  Post dose 3 | 0.03 | 0.06
  Post any dose | 0.30 | 0.51

9. Other Pre Specified Outcome: Serious Adverse Event Assessment
Description: as for outcome 8
Time Frame: After each dose and up to 10 months post-vaccination
Measure: Number; unit: Proportion of participants
Arm/Group | Group A: Standard Dosing | Group B: Alternate Dosing
Number analyzed (Participants) | 33 | 33
Proportion of participants
  Serious Adverse Event-Post dose 1 | 0 | 0
  Serious Adverse Event-Post dose 2 | 0 | 0
  Serious Adverse Event-Post dose 3 | 0.03 | 0

ADVERSE EVENTS:
Time Frame: 7 days after each dose, up to 10 months post-vaccination
Description: Proportions of subjects in each vaccine group reporting a reactogenicity event in the period following each dose and any dose of RV5 will be determined.
Arm/Group | Group A: Standard Dosing | Group B: Alternate Dosing
Serious Adverse Events (participants affected / at risk) | 1/33 | 0/33
Other Adverse Events (participants affected / at risk) | 10/33 | 17/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Standard Dosing (N=33) | Group B: Alternate Dosing (N=33)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Standard Dosing (N=33) | Group B: Alternate Dosing (N=33)
Otitis Media (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear Drainage (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (6) | 8 (10)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 13 (15)
Gastroenteritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Change in stool (Gastrointestinal disorders) | 1 (1) | 4 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestanal upset (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colic (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 4 (4) | 1 (1)
Irritability (General disorders) | 5 (6) | 5 (6)
Poor weight gain (General disorders) | 0 (0) | 1 (1)
Excessive sleepiness (General disorders) | 0 (0) | 1 (1)
Sleeplessness (General disorders) | 0 (0) | 1 (1)
Change in appetite (General disorders) | 0 (0) | 2 (2)
Motor vehicale accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
URI (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Diaper rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Macule on chin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No